CLINICAL TRIAL: NCT01710696
Title: Induction of Puberty With 17-Beta Estradiol in Girls With Turner Syndrome. An Open Randomized Trial
Brief Title: Induction of Puberty With 17-beta Estradiol in Girls With Turner Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHTUR/E/2
Record Dates: First submitted 2012-10-16; First posted 2012-10-19 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Genetic Disorder; Turner Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Turner Syndrome | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual dose (Experimental)
  Interventions: Drug: 17-beta estradiol
- Fixed dose (Experimental)
  Interventions: Drug: 17-beta estradiol

INTERVENTIONS:
Drug: 17-beta estradiol — 5-15 mcg/kg daily for 2 years. Dose readjusted every 3 months. Administered orally
  Arms: Individual dose
Drug: 17-beta estradiol — 0.2 mcg daily for 12 months, dose escalated to 0.5 mcg daily for 12 months. Administered orally
  Arms: Fixed dose

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to induce normal pubertal development in girls with Turner Syndrome in accordance with that of their peers and their individual state psychosocial maturation.

ELIGIBILITY:
Inclusion Criteria:

* Turner Syndrome
* Treatment with growth hormone
* Bone age minimum 12 years and maximum 14 years
* Clear signs of ovarian insufficiency
* Well documented growth rate during the last 12 months

Exclusion Criteria:

* Signs of spontaneous puberty
* Known or suspected hypersensitivity to trial product
* Acute or chronic liver disease
* Previous treatment with estrogen
* Undiagnosed abnormal genital bleeding
* Known thyroid diseases not adeadequately treated
* Porphyria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1998-07-23 (Actual); Primary Completion 2004-07-26 (Actual); Study Completion 2004-07-26 (Actual)

PRIMARY OUTCOMES:
Pubertal stage assesed by Tanner score
FSH (Follicle Stimulating Hormone) levels

SECONDARY OUTCOMES:
Height velocity
Pubertal stage assessed by Tanner score: Breast, pubic hair, axillary hair
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (23):
- Spain (23):
  - Novo Nordisk Investigational Site, Alicante
  - Novo Nordisk Investigational Site, Badajoz
  - Novo Nordisk Investigational Site, Barakaldo
  - Novo Nordisk Investigational Site, Cáceres
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, El Palmar
  - Novo Nordisk Investigational Site, Elche
  - Novo Nordisk Investigational Site, Esplugues Llobregat
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Jaén
  - Novo Nordisk Investigational Site, Las Palmas
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Salamanca
  - Novo Nordisk Investigational Site, San Cristóbal de La Laguna
  - Novo Nordisk Investigational Site, Santa Cruz de Tenerife
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Tarrasa
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Valladolid
  - Novo Nordisk Investigational Site, Zaragoza

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com